CLINICAL TRIAL: NCT00600912
Title: Inflammatory Response and Hepatic Function in Patients Requiring Parenteral Nutrition: Comparison of a Lipid Emulsion Based ob Soybean Oil, Medium-Chain Triglycerides, Olive Oil and Fish Oil Versus a Lipid Emulsion Based on Olive and Soybean Oil
Brief Title: Influence of of a Lipid Emulsion on Inflammatory Response and Hepatic Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Klinikum Ludwigshafen (Other)
Responsible Party: Klinikum Ludwigshafen, Dep. of Anesthesiology, Dr. S. N. Piper
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMOF 5178; kli-Lu-spiper 12-2007
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Inflammatory Response; Hepatic Function
Keywords: lipid emulsion; fish oil; parenteral nutrition; leucotriene LTB5; hepatic function
MeSH Terms: conditions — Hyperphagia | interventions — SMOFlipid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-SMOFlipid® (Experimental): lipid emulsion based on soybean oil, medium-chain triglycerides, olive oil and fish oil SMOFlipid®-Group (n = 21)
  Interventions: Drug: SMOFlipid®
- 2-ClinOleic 20%® (Active Comparator): olive and soybean oil-group (n=21)
  Interventions: Drug: 2-ClinOleic 20%®

INTERVENTIONS:
Drug: SMOFlipid® — continuously, for 5 days postoperatively, corresponding to the observation time. Nonprotein calories: to 60% as glucose and to 40% as lipid emulsion. The total energy intake per day was adjusted to 25 kcal kg-1 body weight.
  Other Names: SMOFlipid 20%® (Fresenius Kabi Deutschland GmbH,Bad Homburg, Germany)
  Arms: 1-SMOFlipid®
Drug: 2-ClinOleic 20%® — continuously, for 5 days postoperatively, corresponding to the observation time. Nonprotein calories: to 60% as glucose and to 40% as lipid emulsion. The total energy intake per day was adjusted to 25 kcal kg-1 body weight.
  Other Names: ClinOleic 20%® (Baxter Deutschland GmbH,Unterschleissheim, Germany)
  Arms: 2-ClinOleic 20%®

SUMMARY:
Lipid emulsions are an essential part of parenteral nutrition, both as a part of energy supply, and as a source of essential fatty acids. It has been shown that the fatty acid composition of cell membranes is influenced by the fatty acid profile of dietary lipids, and may therefore be responsible for modulation of immune response. The aim of this study was to assess the effects of a new lipid emulsion based ob soybean oil, medium-chain triglycerides, olive oil and fish oil compared with a lipid emulsion based on olive and soybean oil on the inflammatory response and hepatic function in postoperative intensive care unit (ICU) patients.

DETAILED DESCRIPTION:
Fatty emulsions are an indispensable part of parenteral nutrition, because they deliver energy and essential fatty acids. Furthermore, lipids are involved in the structure and function of cell membranes and receptors, modifying gene expression, and modulating the inflammatory and immune response. In addition, fatty acids are precursors of prostaglandins and other eicosanoids and have therefore important metabolic functions.A promising substrate in the development of lipid emulsions can be seen in fish oils containing solutions. With regard to the current literature, fish oil have a potential benefical influence on the pathophysiological response to endotoxins and exert important modulations on eicosanoid and cytokine biology.

However, there are no studies avaibale comparing fish oil containing fatty emulsions to a lipid emulsion based on olive and soybean oil with regard to inflammatory response and hepatic function.

Therefore, the aim of this study was to evaluate the effects of a new lipid emulsion based ob soybean oil, medium-chain triglycerides, olive oil and fish oil compared to a lipid emulsion based on olive and soybean oil on the inflammatory response and hepatic function in postoperative intensive care unit (ICU) patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years
* Elective operative procedure, and indication for parenteral nutrition over 5 postoperative days
* ASA I-III
* Haemoglobin > 10 g/dl
* Ability and acceptance to agree to the study participation
* Written informed consent

Exclusion Criteria:

* Liver insufficiency (ASAT, ALAT > 40 U/l)
* Renal insufficiency (creatinine > 1.4 mg/dl)
* Pancreas insufficiency
* Emergencies
* Women in child bearing age and missing negative pregnancy test, pregnancy or lactation
* Diseases from the central nervous system (such as M. Parkinson and multiple sclerosis)
* Alcohol and drug abuse (including opioid abuse)
* Acute pulmonary oedema
* Decompensated cardiac insufficiency
* Insulin-dependent diabetes mellitus
* Overweight (body mass index > 30 kg/m2
* Cachexia (body mass index < 18 kg/m2)
* Psychiatric disorders
* Hypersensitivity to egg, coconut or soy proteins
* Patients taking chronic corticoids
* Allergy to any of the study agents
* Refusal from the patient to participate in the study
* Participation in another study project

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary objective is to monitor the leucotriene (LT) LTB5 in patients requiring parenteral nutrition | 5 days

SECONDARY OUTCOMES:
Hepatic function assessed by measuring alpha-glutathione S-transferase (α-GST), alanin-aminotransferase (ALT),and aspartate-aminotransferase (AST) | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Swen N. Piper, Dr. med., Principal Investigator — Klinikum Ludwigshafen, Department of Anaesthesiology, Ludwigshafen, Germany
Locations (1):
- Klinikum der Stadt Ludwigshafen, Department of Anesthesiology and Intensive Care Medicine, Ludwigshafen, Germany

REFERENCES:
- [Background] Antebi H, Mansoor O, Ferrier C, Tetegan M, Morvan C, Rangaraj J, Alcindor LG. Liver function and plasma antioxidant status in intensive care unit patients requiring total parenteral nutrition: comparison of 2 fat emulsions. JPEN J Parenter Enteral Nutr. 2004 May-Jun;28(3):142-8. doi: 10.1177/0148607104028003142. PMID 15141405
- [Background] Grimm H, Mertes N, Goeters C, Schlotzer E, Mayer K, Grimminger F, Furst P. Improved fatty acid and leukotriene pattern with a novel lipid emulsion in surgical patients. Eur J Nutr. 2006 Feb;45(1):55-60. doi: 10.1007/s00394-005-0573-8. Epub 2005 Jul 22. PMID 16041475
- [Background] Adolph M. Lipid emulsions in parenteral nutrition. Ann Nutr Metab. 1999;43(1):1-13. doi: 10.1159/000012761. PMID 10364625